CLINICAL TRIAL: NCT02928042
Title: Inhibition Effects of Probiotics on Pathogens Associated With Ventilator Associated Pneumonia
Brief Title: Inhibition Effects of Probiotics on Pathogens Associated With VAP
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Collaborators: Dilek Özcengiz (Unknown)
Responsible Party: Principal Investigator, Feride Karacaer, Specialist doctor, Cukurova University
Other Study IDs: PVAP69
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — PrtB protein, bacteria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lactobacillus bacteria: Pseudomonas aeruginosa, Acinetobacter baumanii, Staph aureus and Klebsiella pneumoniae will be isolated from tracheal aspiration cultures. 80 isolates associated with pneumonia will be identified and made antibiogram with VITEK. Then antimicrobial effects of Lactobacillus bacteria (LAB) (Lc. lactis subsp. lactis (IL 1403), Lc. lactis subsp. lactis (ATCC 11454), Lactobacillus plantarum (FI8595), Leuconostoc mesenterodies subsp. cremoris (DSMZ 20346), Streptococcus thermophilus (NCFB2392), Pediococcus acidophilus (ATCC 25741)) and nisin bacteriocin will be investigated on the bacteria's growth rate in the laboratory.
  Interventions: Other: Lactobacillus bacteria

INTERVENTIONS:
Other: Lactobacillus bacteria — Antimicrobial effects of Lactobacillus bacteria (LAB) and nisin bacteriocin on pathogen bacteria and commercial strains of the same bacteria's growth rate will be investigated.

SUMMARY:
This study evaluates that P. aeruginosa, A. baumannii, K. pneumonia and Staph aureus which are obtained from patients' tracheal aspiration culture who treated with mechanical ventilation will be compared with Lactobacillus (LAB) members and nisin bactriocin in the laboratory. The aim is to investigate the probiotics' antimicrobial properties and effects on these bacteria's growth rate.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) is one of the most commonly seen hospital-acquired infections that occurs in patients who receive mechanical ventilation. VAP usually occurs 48-72 hours after mechanical ventilation and is related increased incidence of multidrug-resistant infections, increased antibiotic use, extended mechanical ventilation time, increased patient stay in the intensive care unit (ICU), and increased patient stay in the hospital. One recent intervention is the probiotic therapy which is a nonantibiotic strategy for maintenance of the host's aerodigestive microbial balance and VAP prevention.Common causative pathogens of VAP include Gram negative bacteria such as Pseudomonas aeruginosa, Klebsiella pneumoniae, and Acinetobacter species, and Gram-positive bacteria such as Staphylococcus aureus. In this study, these Gram negative pathogens obtained from mechanical ventilated patients' tracheal aspiration culture and reference bacteria strains will be compared with Lactobacillus (LAB) members and nisin in the laboratory. Probiotics' antimicrobial properties and effects on these bacteria's (obtained from patients and reference strains) growth rate will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who mechanically ventilated at least 48 hours in the intensive care unit

Exclusion Criteria:

* Patients who mechanically ventilated less than 48 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who mechanically ventilated at least 48 hours will be included. Patients' tracheal aspirate cultures will be used for study. Pseudomonas aeruginosa, Acinetobacter baumanii, Staphylococcus aureus and Klebsiella pneumoniae will be isolated from tracheal aspiration cultures.Antimicrobial effects of Lactobacillus members will be investigated on the bacteria's growth rate in the laboratory.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Probiotics' antimicrobial properties and effects on P. aeruginosa, A. baumanii, Staph. auresu and K. pneumonia's growth rate. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Özcengiz, Professor, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandre Y, Le Berre R, Barbier G, Le Blay G. Screening of Lactobacillus spp. for the prevention of Pseudomonas aeruginosa pulmonary infections. BMC Microbiol. 2014 Apr 27;14:107. doi: 10.1186/1471-2180-14-107. PMID 24766663
- [Background] Petrof EO, Dhaliwal R, Manzanares W, Johnstone J, Cook D, Heyland DK. Probiotics in the critically ill: a systematic review of the randomized trial evidence. Crit Care Med. 2012 Dec;40(12):3290-302. doi: 10.1097/CCM.0b013e318260cc33. PMID 22975886